CLINICAL TRIAL: NCT05220215
Title: Compare the Effects of Resistance Band Training and Nordic Hamstring Exercise on Hamstring Strength Among Football Players
Brief Title: Resistance Band Training Versus Nordic Hamstring Exercise on Hamstring Strength Among Football Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/01015 Anas Bin Mujeeb
Record Dates: First submitted 2022-01-03; First posted 2022-02-02 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Intervention; Injury Prevention
Keywords: Nordic Hamstring exercise; Modified sphygmomanometer; Manual muscle Testing; Resistance band

STUDY DESIGN:
Intervention Model Description: Two groups with randomization, Assignment: Nordic Hamstring exercise versus Hamstring Curl with Resistance band
Who Masked: Participant
Masking Description: According to Study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Nordic Hamstring Exercise (Experimental): This group includes 15 male participants who will be given 10 minutes of warm and cool down sessions that includes stretching.
  Number of sets and repetitions progressively increase i-e: Week 1 - 2 sessions with 2 sets of 5 repetitions each. Week 2 - 2 sessions with 3 set of 5 repetitions each. Week 3 - 2 sessions with 4 set of 6 repetitions each. Week 4 - 2 sessions with 4 set of 8 repetitions each.
  Interventions: Other: Nordic Hamstring Exercise
- Group B: Hamstring Curl with Resistance Band (Experimental): This group includes 15 male participants who will be given 10 minutes of warm and cool down sessions that includes stretching.
  Number of sets progressively increase i-e: Week 1 - 2 sessions with 2 sets of 15 repetitions each. Week 2 - 2 sessions with 3 set of 15 repetitions each. Week 3 - 2 sessions with 4 set of 15 repetitions each. Week 4 - 2 sessions with 4 set of 15 repetitions each.
  Interventions: Other: Hamstring Curl with Resistance band

INTERVENTIONS:
Other: Nordic Hamstring Exercise — To perform Nordic Hamstring Exercise, the subject was in kneeling position on the mat, arms by the side or in front of the chest, knee in 90-degree flexion and ankles well stabilized with the help of a therapist which is positioned behind the subject. Then subject was asked to lean forward by using the hamstring muscles by extending while trying to resist the forward fall, he should lean forward from the knee and not from the hip. The only time one can put his hands in front of him is when he can't rely on his legs and then push himself back to starting position and them repeat the procedure again.
  Arms: Group A: Nordic Hamstring Exercise
Other: Hamstring Curl with Resistance band — Traditional Hamstring Curl by using Resistance band.
  Resistance Band: Thera-band Green, 4.6 kg resistance at 100% elongation
  Arms: Group B: Hamstring Curl with Resistance Band

SUMMARY:
The major aim of this project to compare the effects of Resistance band training and Nordic hamstring exercise on hamstring strength among football players.

DETAILED DESCRIPTION:
Hamstring strength is important in football players and plays an important role in their sprint gait cycle. Football players should develop sprinter-like musculature in order to benefit their body strength and power hence preventing from hamstring strain injuries. Professional and recreational sports like Football, hamstring muscle strength training is commonly used to increase and balance lower body strength and power.

ELIGIBILITY:
Inclusion Criteria:

1. Male
2. Age: 18-28 years
3. Football players
4. Playing should be at least for 1 year

Exclusion Criteria:

1. To be involved in any additional strength training program i-e: Gym Activities
2. Athletes having hamstring and Quadriceps injuries
3. History of trauma at knee, hip or back
4. Recent history of any upper and lower extremity fracture
5. Any orthopedic or neurological disorder.

Ages: 18 Years to 28 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 34 (Actual)
Dates: Start 2021-06-29 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Modified sphygmomanometer Test | 4 weeks
  Modified sphygmomanometer is a non-invasive test and method which may provide reliable, rapid and valid measurement of assessing hamstring strength in field-based sports.
Manual Muscle Test (MMT) | 4 weeks
  Manual muscle test (MMT) is a procedure for the evaluation of strength of individual muscle or muscles group, based upon the effective performance of a movement in relation to the forces of gravity or Manual Resistance through the available Range of motion (ROM). Manual Muscle Testing Grading System from 0=No visible or palpable contraction to 5= full range of movement against gravity, maximal resistance.

SECONDARY OUTCOMES:
40-yard dash Test | 4 weeks
  Subjects were asked to be ready in a starting position with the appropriate foot position behind the starting line without any physical movements and subjects ran up to 40-yard when the signal was given out. The stopwatch was started when the players started to run and stopped when they had reached the finishing line. The procedures were repeated for the second time. Two trial results were documented and the best result was taken.
Muscle soreness rating following exercise | 4 weeks
  Participants used a 10-point Numeric Pain Rating scale to record the level of muscle soreness experienced after 1, 2, 4-week training sessions. Ratings of soreness intensity will be assessed consisted of a single 0-10 scale, with "0" indicating "no soreness at all" and "10" indicating the "greatest soreness they could imagine".

CONTACTS AND LOCATIONS:
Overall Officials: Waqar Ahmed Awan, PhD, Principal Investigator — Riphah International University
Locations (1):
- Riphah international university, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monajati A, Larumbe-Zabala E, Goss-Sampson M, Naclerio F. The Effectiveness of Injury Prevention Programs to Modify Risk Factors for Non-Contact Anterior Cruciate Ligament and Hamstring Injuries in Uninjured Team Sports Athletes: A Systematic Review. PLoS One. 2016 May 12;11(5):e0155272. doi: 10.1371/journal.pone.0155272. eCollection 2016. PMID 27171282
- [Background] Mjolsnes R, Arnason A, Osthagen T, Raastad T, Bahr R. A 10-week randomized trial comparing eccentric vs. concentric hamstring strength training in well-trained soccer players. Scand J Med Sci Sports. 2004 Oct;14(5):311-7. doi: 10.1046/j.1600-0838.2003.367.x. PMID 15387805
- [Background] Rey E, Paz-Dominguez A, Porcel-Almendral D, Paredes-Hernandez V, Barcala-Furelos R, Abelairas-Gomez C. Effects of a 10-Week Nordic Hamstring Exercise and Russian Belt Training on Posterior Lower-Limb Muscle Strength in Elite Junior Soccer Players. J Strength Cond Res. 2017 May;31(5):1198-1205. doi: 10.1519/JSC.0000000000001579. PMID 27467517
- [Background] Huggins, S, Davies, N, Evans, KL, and Williams, MD. Nordic hamstring exercise strength changes over a season in academy footballers. Br J Sports Med. 2017; 51: 332.
- [Background] Babu SK, Paul A. Effectiveness of Nordic hamstring exercise in improving hamstring muscle flexibility, strength and endurance among young adults. Int J Health Sci Res. 2018; 8(3):119-132